CLINICAL TRIAL: NCT04056793
Title: A Qualitative Study to Assess the Feasibility and Acceptability of an Optimized Birthing Position
Brief Title: Acceptability Assessment of an Optimized Birthing Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, DAVID DESSEAUVE, Médecin cadre - MD, PhD, PD-MER, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-00872
Record Dates: First submitted 2019-08-09; First posted 2019-08-14 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Birth; Prolonged
Keywords: Birthing position; Dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parturients in situation of dystocia (Experimental): Positioning of the parturients in an optimized birthing position
  Interventions: Other: Optimized birthing position

INTERVENTIONS:
Other: Optimized birthing position — The parturients will be asked to adopt a supine position with a hyperflexion of the thighs and a flat back, and to maintain the position for a duration of twenty minutes.

SUMMARY:
This qualitative study evaluates the acceptability of positioning pregnant women in labour in an optimized position, which consists in the hyperflexion of the legs and the loss of the lumbar lordosis. Twenty patients in situation of dystocia will adopt the described position for a limited amount of time.

DETAILED DESCRIPTION:
Recent data brings out that the Caesarian Section rate in Switzerland is quite high, reaching 33.4 %. Though, the reasons to this increasing amount of CS are not fully known. Therefore, it is absolutely necessary to expand the existing knowledge in different fields, including the biomechanics of childbirth. Numerous CS are performed in response to an obstructed labour, especially when the foetus does not engage in the pelvis near full dilatation. In order to manage such situations, midwifes currently position parturients in pragmatic postures. Although not verified by data, this care management suggests that it is possible to impact the position of the bone segments at stake for vaginal birth including pelvis and lumbar spine and to promote the descent of the foetus through the pelvic inlet plane. In his PhD thesis about vaginal birth biomechanics, Desseauve et al investigated this area and found out that an optimized position similar to the squatting position (hyperflexion of the thighs and loss of the lumbar lordosis) could be close to the perfect delivery position in terms of ability for the foetus to go through the pelvic inlet plane. Although these findings are encouraging, it is yet to be confirmed in clinical practice, particularly when a dystocia occurs. Prior to doing that, it is though necessary to validate the optimized posture in terms of acceptability in a qualitative clinical study. In this study, fifteen to twenty parturients who respond to the inclusion criteria and whose foetus does not engage in the pelvis near full dilation will be asked to adopt the optimized position for a twenty minutes period. The investigator will then consign information reflecting the progress of the labour on a data sheet.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* Parturient in situation of mechanical dystocia (non engagement at full dilation)

Exclusion Criteria:

* Inability or medical contraindications to undergo the investigated intervention (e.g. orthopaedic injury or disease preventing the parturient from adopting the optimised position)
* Clinically significant concomitant diseases
* Incapacity of judgment
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia, etc.
* Foetus cardiac rhythm disorder

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the optimized birthing position assessed by calculating the average score obtained through the VAS | 20 minutes
  The Visual Analogue Scale will allow to obtain a score from 0 to 10, 0 standing for complete dissatisfaction and 10 for complete satisfaction of the participants

SECONDARY OUTCOMES:
Number of refusals | 20 minutes
  Number of parturients who will refuse to participate to the study
Number of risk factors of non-engagement of the foetus at full dilation | 20 minutes
  The risk factors are constituted of macrosomy, medical induction of labour, artificial rupture of membranes, hypokinesia (<5 uterine contractions/min), use of oxytocin and presence of a peridural anaesthesia
Neonatal adaptation assessed by the Apgar score | 20 minutes
  The Apgar score will be evaluated at 1, 5 and 10 minutes
Birth outcome assessed by the percentage of vaginal delivery, Caesarian Section, delivery hemorrhage and perineal tear | 20 minutes
Weight of the foetus measured in kilograms | 20 minutes
Height and head circumference of the foetus measured in centimeters | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pr David Baud - Médecin chef de service - MD, PHD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No